CLINICAL TRIAL: NCT04036929
Title: Hand Osteoarthritis: Investigating Pain Effects in a Randomised Placebo-controlled Feasibility Study of an Estrogen-containing Therapy
Brief Title: Can we Use Estrogen-containing Therapy to Improve Pain in Women After Menopause With Hand Osteoarthritis?
Acronym: HOPE-e
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Oxford Clinical Trials Research Unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HOPE-e
Record Dates: First submitted 2019-06-21; First posted 2019-07-30 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Hand Osteoarthritis
Keywords: Osteoarthritis; Hand; Hormone; Pain; Estrogen
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Estrogen-bazedoxifene (Experimental): Tablet, once daily for 6 months.
  Interventions: Drug: Estrogen-bazedoxifene
- Placebo (Placebo Comparator): Closely matched tablet, once daily for 6 months.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Estrogen-bazedoxifene — Conjugated estrogens 0.45 mg-bazedoxifene acetate 20 mg.
  Other Names: Duavive
  Arms: Estrogen-bazedoxifene
Drug: Placebo oral tablet — Placebo oral tablet
  Arms: Placebo

SUMMARY:
Post-menopausal women aged 40-65 with symptomatic hand osteoarthritis are invited to take part in this feasibility study. The study's aim is to investigate whether it is acceptable to women with painful hand OA to take an estrogen-containing therapy, and what is the best way of collecting some of the information in order to facilitate planning a full size trial. The investigator's long-term aim is to find out whether giving estrogen-containing therapy to women after the menopause improves hand OA symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed written consent
* Female, aged 40-65 years old
* In those with an intact uterus: At least 12 months of spontaneous amenorrhea (without any menstrual bleeding in last 12 months) and last menstrual period not more than 10 years ago
* In those who have undergone hysterectomy or are/were using an intrauterine contraceptive device with progesterone local therapy (such as Mirena): Follicle stimulating hormone (FSH) ≥30 milli-International Units per millilitre (mIU/ml) on screening blood test AND a history of menopausal symptoms in the last 1 to 10 years, in keeping with appropriate timing of menopausal status
* Hand pain, aching or stiffness on most days in the last 3 months
* At least 2, painful hand joints of any type (interphalangeal joints (IPJ) or base of thumbs)
* Fulfils American College of Rheumatology clinical diagnostic criteria for hand OA (3 or more of following):

  1. Hard tissue enlargement of 2 or more of the following joints: 2nd or 3rd distal interphalangeal joints (DIPJ), 2nd or 3rd proximal interphalangeal joints (PIPJ), first carpometacarpal joints (CMCJ)
  2. Hard tissue enlargement of 2 or more of the DIPJs
  3. Less than 3 swollen metacarpophalangeal joints (MCPJ)
  4. Deformity of at least one of the joints listed in first point

OR, for those with base of thumb osteoarthritis only not fulfilling these criteria, has clinical symptoms and examination findings consistent with base of thumb osteoarthritis.

* Hand pain has not responded adequately to National Institute for Health and Care Excellence core guidance for management of OA, including the use of paracetamol or non-steroidal anti-inflammatory drug (NSAID) gel, except where there is contraindication or intolerance
* Average hand pain is reported as typically more than 4 out of 10 in severity, or average hand pain in the last 7 days of 4/10 or more on a visual analogue scale
* In the Investigator's opinion, is able and willing to comply with all study requirements

Exclusion criteria

* Other cause of hand pain, including inflammatory arthritis, connective tissue disorder, chronic pain or alternative clinical diagnosis such as tenosynovitis or carpal tunnel syndrome
* Pregnancy or breast feeding, or risk of this during study
* Use of one or more prohibited treatments within specified timeframe, or not willing to avoid treatment for the duration of the study:

  * Oral contraceptive pill, or systemic HRT within the last 6 months (Use of an intrauterine contraceptive device with progesterone local therapy (Mirena) or vaginal topical estrogen use (known low systemic absorption) are not exclusions to participation)
  * Anti-estrogen medication within the last 6 months
  * Oral, intramuscular or intraarticular steroid within the last 3 months
  * Intraarticular hyaluronan to a hand joint within the last 6 months
  * Initiation of new oral analgesia within the last 4 weeks
  * Initiation of glucosamine, chondroitin, hand exercises or other relevant non- pharmacological therapy within the last 6 weeks
  * Hand surgery within the last 6 months, or planned within the next 6 months
  * Medications likely to increase hepatic metabolism of study medication, including:
  * St. John's Wort
  * Anti-convulsants (phenobarbital, phenytoin, carbamazepine, lamotrigine)
  * Some anti-infectives (rifampicin, rifabutin, nevirapine, efavirenz, ritonavir and nelfinavir)
* Presence of one or more medical contraindications to the use of systemic hormonal replacement therapy:

  * In those aged 40-45 years, FSH <30 mIU/ml on screening blood test, i.e. non- confirmatory of menopausal status
  * Any history of breast, endometrial, ovarian or skin cancer
  * Any other history of other cancer within 5 years (except treated Basal Cell Carcinoma, BCC)
  * Relevant breast issue on routine national breast screening in prior 3 years
  * Undiagnosed genital bleeding, or untreated endometrial hyperplasia, active uterine fibroids or endometriosis
  * Active or past history of venous thromboembolism (VTE) (including deep venous thrombosis, pulmonary embolism and retinal vein thrombosis), or at high risk of VTE (such as known thrombophilic disorders (such as Protein C, S or anti-thrombin deficiency) or presence of a strong family history of VTE). Women with a first degree relative with a history of VTE, or other strong family history of VTE at the Investigators' discretion.
  * Active or past history of arterial thrombo-embolic disease (such as myocardial infarction, angina or stroke) or strong family history of stroke)
  * Clinically significant immobility
  * Migraine or active epilepsy
  * Uncontrolled hypertension (or diastolic pressure greater than 90 mmHg or systolic pressure greater than 145 mmHg at screening visit)
  * Uncontrolled diabetes mellitus or uncontrolled hypertriglyceridaemia
  * Body Mass Index (BMI) greater than 30
  * Active malabsorption syndrome or clinically significant small bowel disease
  * Acute liver disease, clinically significant abnormal liver function, active gallbladder disease or porphyria
  * Clinically significant renal impairment
  * Intolerance to lactose, fructose or glucose (including galactose intolerance, lactase deficiency, fructose intolerance, glucose-galactose malabsorption or sucrase- isomaltase insufficiency)
  * Known sensitivity to either conjugated equine estrogens, bazedoxifene or the combination
* Any other significant or uncontrolled disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study
* Participants who have participated in another research trial involving an investigational product in the past 8 weeks

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Feasibility: Rates of eligible participant identification, rates of recruitment/randomisation from different sources, retention rates | From the date of recruitment opening until the date of recruitment closing, 1 year
Feasibility: Frequency of adverse events related to the active study medication | Through study completion, 7 months
Feasibility: Bang's Blinding Index (likelihood of unblinding) | Week 24
  Self-complete questionnaire which assesses likelihood that participant or Investigator have become unblinded
Feasibility: Monitoring study medication compliance (via diaries) | From randomisation to end of treatment at Week 24
  Participants will be asked to record any missed doses of study medication on a paper diary which will be provided at each visit. We will ask participants to bring the diary to each study visit and any missed doses will be recorded in the Case Report Form.

SECONDARY OUTCOMES:
Pain and function: Average hand pain over last 14 days (NRS 0-10) | Collected at: Baseline, Week 4, Week 12, Week 24
  Numerical Rating Scale 0-to-10, where 0 is "no pain" and 10 is "pain as bad as you can imagine"
Pain and function: Remote pain-rating prior to a visit (NRS 0-10) | Collected at: Baseline, Week 4, Week 12, Week 24
  Numerical Rating Scale 0-to-10, where 0 is "no pain" and 10 is "pain as bad as you can imagine"
Pain and function: Prevalence of joint pain elsewhere (pain manikin) | Collected at: Baseline, Week 12, Week 24
  Prevalence of joint pain elsewhere in the 4 weeks preceding the study visit
Pain and function: Functional Index for Hand OA (FIHOA) | Collected at: Baseline, Week 12, Week 24
  Validated measurement of hand OA-related functional impairment. It includes 10 questions scored according to a 4-grade scale. The score ranges from 0 (no functional impairment) to 30 points (maximal impairment).
Pain and function: EQ-5D-5L | Collected at: Baseline, Week 12, Week 24
  Validated measurement of quality of life across five dimensions and their associated levels of severity on a 1 (no problems) to 5 (extreme problems) scale.
Menopause symptoms: The Menopause Specific Quality of Life Questionnaire (MENQOL) | Collected at: Baseline, Week 12, Week 24
  Validated measurement of menopausal symptoms and their associated degree of severity; 30 items in a Likert-scale format. Items are rated as present or not present and if present how bothersome, on a 0 (not bothersome) to 6 (extremely bothersome) scale.
  The interventional version is being used here, which includes an additional 3 questions relevant to Hormonal Replacement Therapy (HRT) use which has been used in a trials setting.
Menopause symptoms: Greene Climacteric Scale | Collected at: Baseline, Week 12, Week 24
  A 21-item validated questionnaire that measures a variety of menopausal symptoms on a 4-point Likert scale (0 = "not at all" to 3 = "extremely"), plus one sexual function probe.
Joint appearance: Cosmesis score of Michigan Hand Questionnaire (4 questions, questions 28-31) | Collected at: Baseline, Week 12, Week 24
  Subdomain of hand-specific outcomes instrument that measures outcomes of patients with conditions of, or injury to, the hand or wrist.
Joint appearance: Investigator-recorded tender and swollen joint counts | Collected at: Baseline, Week 12, Week 24
  Investigator examination of tender and swollen hand joints, binary recording (1 swollen, 0 not swollen).
Joint appearance: Photographic recording of swollen hand joints | Collected at: Baseline, Week 12, Week 24
  Standardised digital photography of hands
Joint function: Jamar grip strength - average of 3 measurements | Collected at: Baseline, Week 12, Week 24
  Handgrip strength will be measured in kilograms to the nearest hundred grams in both hands using a Jamar dynamometer.
  Both hands will be alternately assessed three times and the average score recorded.
End of Treatment questionnaire (study-specific) | Week 24
  A study specific end of treatment questionnaire will be designed to include items on acceptability.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - White Horse Medical Practice, Faringdon Medical Centre, Faringdon, Oxfordshire
  - Charing Cross Hospital, Imperial College Healthcare NHS Trust, London
  - Nuffield Orthopaedic Centre, Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No
Access to the de-identified dataset for purposes of research other than this study, would be at the discretion of the Chief Investigator, Dr Fiona Watt and OCTRU. All participants have consented to the information collected about them from the study may be used in a de-identified form to support other research on hand osteoarthritis in the future and may in certain circumstances be passed on to other collaborators of the research team in organisations other than the University of Oxford, which may include those outside the EU and commercial organisations. Requests for the de-identified dataset generated during the current study should be made to the Chief Investigator, Dr Fiona Watt (fiona.watt@kennedy.ox.ac.uk) or OCTRU (octrutrialshub@ndorms.ox.ac.uk). Dr Fiona Watt and OCTRU will consider requests once the main results from the study have been published up until 10 Dec 2036 . All requests must relate to bone fide research into hand osteoarthritis research.

REFERENCES:
- [Background] Marian IR, Goff M, Williams JAE, Gulati M, Chester-Jones M, Francis A, Watson M, Vincent TL, Woollacott S, Mackworth-Young C, Glover V, Furniss D, Gardiner M, Lamb SE, Vincent K, Barber VS, Black J, Dutton SJ, Watt FE. Hand Osteoarthritis: investigating Pain Effects of estrogen-containing therapy (HOPE-e): a protocol for a feasibility randomised placebo-controlled trial. Pilot Feasibility Stud. 2021 Jun 24;7(1):133. doi: 10.1186/s40814-021-00869-1. PMID 34167594
- See also: HOPE-e study website — https://hope.octru.ox.ac.uk/